CLINICAL TRIAL: NCT04425811
Title: The Effect of Kinesiological Taping Applied to the Tibialis Anterior Muscle on Gait Parameter in Stroke Patients: Sham Controlled Study
Brief Title: The Effect of Kinesiological Taping Applied to the Tibialis Anterior Muscle on Gait Parameter in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Muammer Çorum, Lecturer, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: pamukkaleU
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: Stroke; Kinesiological Taping; Walking; Tibialis Anterior
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Sham Controlled Study
Who Masked: Participant
Masking Description: Original kinesiological tape was applied to the participants. Then sham banding application was done with sticking plaster tape.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No tape applied (No Intervention): Walking parameters were evaluated without any intervention.
- Kinesiological Tape (Experimental): Walking parameters were evaluated after kinesiological taping on the tibialis anterior muscle
  Interventions: Other: kinesiological taping
- Sham taping (Sham Comparator): Walking parameters were evaluated after sham taping on the tibialis anterior muscle
  Interventions: Other: kinesiological taping

INTERVENTIONS:
Other: kinesiological taping — The kinesiological banding applied to the tibialis anterior muscle was applied to improve walking parameters and compared to sham control.
  Arms: Kinesiological Tape; Sham taping

SUMMARY:
The effect of kinesiological taping applied to the tibialis anterior muscle on gait parameter in stroke patients: Sham controlled study

DETAILED DESCRIPTION:
Objective: The aim of this study was to compare the immediate effect of kinesiological and / or sham taping to the tibialis anterior muscle on walking parameters in stroke individuals.

Methods: The study included 28 adults stroke patients . The subjects who received scores of 7 or more in the Hodkinson Mental Test and 3 and above in the Functional Ambulation Classification with subjects who gastrocnemius muscle spasticity 2 and below points according to Modified Ashworth Scale were included in the study. The walking parameters of the participants were evaluated with the BTS G-Walk Spatio-Temporal Walking Analysis System. The walking parameters of the participants who were selected by randomization method were evaluated separately by applying kinesiological taping and sham taping or without any taping or interference on a 10 meter track.

ELIGIBILITY:
Inclusion Criteria:

* 28 stroke individuals (hemiplegic / hemiparetic) who were treated in the Adult
* Neurological Rehabilitation Unit of Pamukkale University Medical Faculty Hospital were included in the study.
* Being between the ages of 25-70
* Volunteers with written consent
* With a 1-year history of stroke
* Who had a stroke for the first time
* Having a lesion in one brain hemisphere

Exclusion Criteria:

* Having neurological or orthopedic comorbid disease
* Patients with a gastrocnemius spasticity greater than 2 according to the modified ashworth scale
* Patients with communication problems
* Patients with cognitive functions below 7 points according to the Hodkinson Mental Test
* Patients with ambulation level below 3 according to Functional Ambulation Classification

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
non-taping walking parameter measurement | 2 hours
  The dominant side lower extremity of the participants was determined as the first preferred lower limb to take steps when walking. Walking parameters of the participants included in the study were evaluated with BTS G-Walk Spatio-Temporal Gait Analysis System. Before the banding applications of the patients, walking parameters were measured by asking them to walk with a shoe that they always use daily with the command "walk normally" on a 10-meter course, and stop with the command "stop" after 10 meters.

SECONDARY OUTCOMES:
With kinesiological taping walking parameter measurement | 2 hours
  Kinesiological taping or sham taping was performed by a certified physiotherapist 2 hours after the measurement of walking parameters without any intervention. Kinesiological banding for the tibialis anterior muscle was performed using muscle technique (stimulation). The taping was performed with the patients lying on a stretcher in the supine position. The kinesiological band was cut in the shape of I considering the participant's muscle length, the edges were ovalized, and the skin was purified from moisture, hair and oil. While applying the muscle technique (stimulation), the tibialis anterior muscle was stretched in the plantar flexion and eversion position. It was then activated by applying heat along the band. After the band was activated, the walking parameters of the participant were measured again with the BTS G-Walk device.
With sham taping walking parameter measurement | 2 hours
  The sham taping was applied to the participants a week or a week before the application of the kinesiological tape. Sham taping application was applied to the same area as kinesiological taping application, but no technique was used. After the Sahm taping application, the walking parameters of the participants were measured again with the BTS G-Wlak device.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Baskan, Phd, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No